CLINICAL TRIAL: NCT00256724
Title: Evaluation of an Inspiratory Impedance Threshold Device (ITD) in the Emergency Department for the Treatment of Hypotension
Brief Title: Efficacy Study of a Facemask Device to Treat Hypotension
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Advanced Circulatory Systems (Industry)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 43-0278-00; Contract W81XWH-04-C-0022
Record Dates: First submitted 2005-11-18; First posted 2005-11-22 (Estimated); Results first posted 2013-07-18 (Estimated); Last update posted 2013-07-31 (Estimated); Status verified 2013-07

CONDITIONS: Hypotension
Keywords: hypotension; hypovolemia; dehydration; sepsis; blood loss
MeSH Terms: conditions — Hypotension; Hypovolemia; Dehydration; Sepsis; Hemorrhage

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sham ITD (Sham Comparator): sham Impedance Threshold Device
  Interventions: Device: sham ITD
- active ITD (Active Comparator): active impedance threshold device
  Interventions: Device: Impedance Threshold Device

INTERVENTIONS:
Device: Impedance Threshold Device — Active impedance threshold device
  Other Names: ResQGard
  Arms: active ITD
Device: sham ITD — sham impedance threshold device
  Arms: Sham ITD

SUMMARY:
The purpose of this study is to determine if the impedance threshold device (ITD) attached to a facemask can increase blood pressure in patients who present to the emergency department with hypotension secondary to hypovolemia. The cause of hypovolemia could be blood loss, sepsis, or dehydration.

DETAILED DESCRIPTION:
The study is designed to test the hypothesis that use of the ITD will result in a rapid rise in blood pressure secondary to an increase in cardiac output. Either an active or sham ITD will be applied to hypotensive patients when initially presented to the emergency department with a systolic blood pressure of <95mmHg. The main endpoint of this study will be the rise in blood pressure over the first 10 minutes of use. Based upon pre-clinical studies as well as clinical studies performed to date, we hypothesize that use of the active ITD will result in a more rapid and higher blood pressure than the sham ITD. Multiple additional clinical parameters will also be compared between the two groups of patients.

ELIGIBILITY:
Inclusion Criteria:

* Conscious patient
* Systolic blood pressure < 95 mmHg
* Hypotension caused by blood loss, sepsis, or dehydration

Exclusion Criteria:

* Hypotension secondary to heart failure
* Complaints of chest pain
* History of heart failure
* Complaints of shortness of breath

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2005-06; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Keith Lurie, MD, Principal Investigator — Advanced Circulatory Systems
Locations (1):
- Hennepin County Medical Center, Minneapolis, Minnesota, United States

REFERENCES:
- [Background] Convertino VA, Cooke WH, Lurie KG. Inspiratory resistance as a potential treatment for orthostatic intolerance and hemorrhagic shock. Aviat Space Environ Med. 2005 Apr;76(4):319-25. PMID 15828629
- [Background] Convertino VA, Ratliff DA, Crissey J, Doerr DF, Idris AH, Lurie KG. Effects of inspiratory impedance on hemodynamic responses to a squat-stand test in human volunteers: implications for treatment of orthostatic hypotension. Eur J Appl Physiol. 2005 Jul;94(4):392-9. doi: 10.1007/s00421-005-1344-1. Epub 2005 Apr 28. PMID 15864634
- [Background] Convertino VA, Ratliff DA, Ryan KL, Doerr DF, Ludwig DA, Muniz GW, Britton DL, Clah SD, Fernald KB, Ruiz AF, Lurie KG, Idris AH. Hemodynamics associated with breathing through an inspiratory impedance threshold device in human volunteers. Crit Care Med. 2004 Sep;32(9 Suppl):S381-6. doi: 10.1097/01.ccm.0000134348.69165.15. PMID 15508665
- [Result] Smith SW, Parquette B, Lindstrom D, Metzger AK, Kopitzke J, Clinton J. An impedance threshold device increases blood pressure in hypotensive patients. J Emerg Med. 2011 Nov;41(5):549-58. doi: 10.1016/j.jemermed.2010.05.013. Epub 2010 Jul 15. PMID 20634018
- See also: Advanced Circulatory Systems, Inc. home page — http://www.advancedcirculatory.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from the emergency department based on age (18-85)and systolic blood pressure ≤95mmHg who were conscious and presumed to have hypotension due to hypoivolemia or relative hypovolemia (blood loss, dehydration, or sepsis).
Period: Overall Study
Arm/Group | Sham ITD | Active ITD
Started | 23 | 24
Completed | 18 | 16
Not Completed | 5 | 8
Not completed — Physician Decision | 2 | 5
Not completed — Protocol Violation | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sham ITD | Active ITD | Total
Number analyzed (Participants) | 23 | 24 | 47
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 1 | 1
  Between 18 and 65 years | 20 | 20 | 40
  >=65 years | 3 | 3 | 6
Age Continuous [Mean (Standard Deviation); unit: years] | 51.6 (11.8) | 46.8 (17.3) | 49.1 (15.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 15 | 28
  Male | 10 | 9 | 19
Region of Enrollment [Number; unit: participants]
  United States | 23 | 24 | 47

OUTCOME MEASURES:

1. Primary Outcome: Rise in Systolic Blood Pressure Over the First 10 Minutes of Use Compared to Baseline
Time Frame: every 2 minutes during 10 minutes of device use
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Sham ITD | Active ITD
Number analyzed (Participants) | 18 | 16
mm Hg | 5.9 (5.9) | 12.9 (8.5)

2. Secondary Outcome: Quantity of Fluid Administration
Time Frame: during 10 minutes of device use
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Sham ITD | Active ITD
Number analyzed (Participants) | 18 | 16
mL | 175 (197) | 93 (170)

ADVERSE EVENTS:
Arm/Group | Sham ITD | Active ITD
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/24
Other Adverse Events (participants affected / at risk) | 0/23 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No